CLINICAL TRIAL: NCT00705263
Title: Evaluation of Satisfaction in Patients Receiving PegIntron Pen/Rebetol for Hepatitis C in Slovenia
Brief Title: Satisfaction in Patients Receiving the PegIntron Pen Plus Rebetol for Hepatitis C (Study P04244)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Schering-Plough (Industry)
Responsible Party: Head, Clinical Trials Registry & Results Disclosure Group, Schering-Plough
Other Study IDs: P04244
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Hepatitis C, Chronic; Hepacivirus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis C: Patients with chronic hepatitis C who are treated with the PegIntron pen plus Rebetol will answer questions on the patient questionnaire.
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b and ribavirin will be administered according to the products' labeling.
  Other Names: PegIntron, PegPen
Drug: Ribavirin (SCH 18908) — Peginterferon alfa-2b and ribavirin will be administered according to the products' labeling.
  Other Names: Rebetol

SUMMARY:
The current gold standard for treatment of chronic hepatitis C is pegylated interferon plus ribavirin. Drug administration accuracy and ease of use will definitely determine treatment effectiveness. This is the idea behind the development and usage of the PegIntron pen (PegPen). Therefore, it is worthwhile to evaluate patients' satisfaction with this novel device. The results of the study will be used to improve PegPen training techniques for patients and health care providers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C treated with the PegIntron pen plus Rebetol

Exclusion Criteria:

* Not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C treated with the PegIntron pen plus Rebetol at sites in Slovenia.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 113 patients were enrolled in the study; however, data were available for 110 subjects
Period: Overall Study
Arm/Group | Patients With Chronic Hepatitis C
Started | 110 (113 patients started the treatment; however, data were available for only 110 patients.)
Completed | 108
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Chronic Hepatitis C
Number analyzed (Participants) | 110
Age Continuous [Mean (Standard Deviation); unit: years] | 40.25 (12.71)
Sex/Gender, Customized [Number; unit: participants]
  Female | 37
  Male | 68
  Not provided | 5
Region of Enrollment [Number; unit: participants]
  Slovenia | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Satisfied With the PegIntron Pen, Including the Assessment of the Device Accuracy and Ease of Use.
Description: Participants were asked to evaluate the training they received in the proper use of the pen, the preparation and injection of the medicine, and to provide their subjective impressions about the use of the PegIntron pen. Satisfaction was defined as score 5 or above on a 7-point grading scale.
Time Frame: After 4 weeks of treatment.
Population: Patients with chronic hepatitis C treated with PegIntron pen plus Rebetol
Measure: Number; unit: Satisfied Participants
Arm/Group | Patients Treated With PegIntron Pen Plus Rebetol
Number analyzed (Participants) | 110
Satisfied Participants
  Injection technique: correctly injected | 104
  No difficulties injecting | 102
  Overall impression | 102
  Satisfaction with the pen | 102
  Ease of setting the dose | 101
  Ease of use of the pen | 101
  Convenience of use of the pen | 101
  Easy injection | 98
  Correct dose | 98
  Helpfulness of the brochure: instructions | 96
  Overall helpfullness of the brochure | 94
  Helpfulness of the brochure: advice | 91
  Helpfulness of the brochure: general information | 90
  Difficulty of preparing the pen | 90
  Time required to prepare the pen | 88

ADVERSE EVENTS:
Arm/Group | Patients With Chronic Hepatitis C
Serious Adverse Events (participants affected / at risk) | 0
Other Adverse Events (participants affected / at risk) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less